CLINICAL TRIAL: NCT02061540
Title: A Pilot, Open-Label Study to Evaluate the Safety, Tolerability and Efficacy of LUM001, an Apical Sodium-dependent Bile Acid Transporter Inhibitor (ASBTi), in Patients With Primary Sclerosing Cholangitis
Brief Title: Open Label Study to Evaluate Safety and Efficacy of LUM001 in Patients With Primary Sclerosing Cholangitis
Acronym: CAMEO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM001-401; 2014-005558-21 (EudraCT Number)
Record Dates: First submitted 2014-02-11; First posted 2014-02-13 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Primary Sclerosing Cholangitis (PSC)
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LUM001 (Experimental): LUM001 administered orally once each day
  Interventions: Drug: LUM001

INTERVENTIONS:
Drug: LUM001 — LUM001 oral dose

SUMMARY:
The study is an open-label study in adults with primary sclerosing cholangitis to evaluate the safety, tolerability, and effect of 14-weeks of daily dosing of LUM001.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between the ages of 18-80 years, inclusive.
2. Diagnosis of PSC
3. If inflammatory bowel disease (IBD) is present, disease activity ≤ 2 (normal to moderate), using the physician assessment on the Mayo ulcerative colitis (UC) disease activity score.
4. Patients receiving azathioprine for intestinal bowel disease are eligible to participate in the study provided that they have had no IBD exacerbations for at least 6 months.
5. Females of childbearing potential must have a negative serum pregnancy test [β human chorionic gonadotropin (β-hCG)] during screening and negative urine pregnancy test at the baseline/Day 0 visit.
6. Sexually active females must be postmenopausal, surgically sterile, or if premenopausal, be prepared to use an effective method (≤ 1% failure rate) of contraception during the trial.
7. Ability to read and understand English in order to use the study-related questionnaires and the text on the eDiary screen.
8. Must be willing and able to use an eDiary daily for a minimum of 20 weeks.
9. Must digitally accept the licensing agreement in the eDiary software at the outset of the study.
10. Must complete at least 10 eDiary Adult ItchRO reports (AM or PM) during each of two consecutive weeks of the screening period prior to allocation to treatment (maximum possible reports = 14 per week).
11. Access to phone for scheduled calls from study site.
12. Must agree to comply with the study protocol procedures and provide written informed consent.

Exclusion Criteria:

1. Small duct PSC (clinical biochemical and histological features compatible with PSC, but having a normal cholangiogram).
2. Presence of a dominant stricture unless brushings and/or biopsies of the stricture are negative for dysplasia or malignancy within 6 months of screening.
3. Surgical or endoscopic biliary tree interventions for treatment of clinically significant strictures within 6 months of screening.
4. IBD flare (Mayo UC disease activity score > 5 including endoscopic evaluation) within 3 months prior to screening.
5. Secondary cause of sclerosing cholangitis (e.g., choledocholithiasis, post-surgical biliary stricture, intra-arterial chemotherapy, recurrent pancreatitis, IgG4 associated cholangiopathy, AIDS cholangiopathy).
6. AST or ALT ≥ 5 x ULN at screening.
7. History or presence of any other concomitant significant liver disease as assessed by the Investigator.
8. Medical conditions that may cause nonhepatic increases in ALP (e.g., Paget's disease).
9. Known history of human immunodeficiency virus (HIV) infection.
10. The anticipated need for a surgical procedure within 20 weeks from randomization.
11. Any female who is pregnant or lactating or who is planning to become pregnant within 20 weeks of randomization.
12. History of cancer, except for basal or squamous cell carcinoma of the skin, or with any laboratory or physical exam or diagnostic procedure finding suggestive of current malignancy.
13. Family history of any documented hereditary cancer syndrome.
14. History of alcohol or other substance abuse within 1 year prior to screening.
15. Receipt of an investigational drug, biologic, or medical device within 30 days prior to Screening, or 5 half-lives of the study agent, whichever is longer.
16. History of noncompliance with medical regimens, unreliability, mental instability or incompetence that could compromise the validity of informed consent or lead to noncompliance with the study protocol.
17. Any other conditions or abnormalities which, in the opinion of the Investigator or Medical Monitor, may compromise the safety of the subject, or interfere with the subject participating in or completing the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Mirum
Locations (9):
- United States (5):
  - Scripps Clinic, La Jolla, California
  - University of California at Davis, Sacramento, California
  - University of Colorado, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Duke University, Durham, North Carolina
- Canada (2):
  - University of Calgary Liver Unit, Calgary, Alberta
  - University Health Network, Toronto Western Hospital, Toronto, Ontario
- United Kingdom (2):
  - University of Birmingham, Birmingham, England
  - Royal Free Hospital, London

REFERENCES:
- [Derived] Bowlus CL, Eksteen B, Cheung AC, Thorburn D, Moylan CA, Pockros PJ, Forman LM, Dorenbaum A, Hirschfield GM, Kennedy C, Jaecklin T, McKibben A, Chien E, Baek M, Vig P, Levy C. Safety, tolerability, and efficacy of maralixibat in adults with primary sclerosing cholangitis: Open-label pilot study. Hepatol Commun. 2023 May 15;7(6):e0153. doi: 10.1097/HC9.0000000000000153. eCollection 2023 Jun 1. PMID 37184523

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 8 centers in Great Britain, Canada, and the United States between 22 April 2014 and 12 February 2016.
Pre-assignment Details: A total of 37 participants were screened, of them 27 participants were enrolled in the study.
Groups:
- Maralixibat (LUM001): Participants received LUM001 tablet orally once daily at a dose of 0.5 milligram (mg) during Week 1; 1 mg during Week 2; 2.5 mg during Week 3; 5 mg during Week 4; 7.5 mg during Week 5; 10 mg during Week 6 followed by stable dosing of 10 mg for 8 weeks.
Period: Overall Study
Arm/Group | Maralixibat (LUM001)
Started | 27
Down-Titrated on LUM001 During the Study | 5
Completed | 23
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of the investigational product.
Arm/Group | Maralixibat (LUM001)
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.7 (11.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) was defined as any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE was considered to be related to the investigational drug product. TEAEs were AEs with a start date on or after the first dose of investigational product and started prior to the last dose of investigational product plus 14 days.
Time Frame: From start of study drug administration until Week 18
Population: Safety population included all participants who received at least 1 dose of the investigational product.
Measure: Number; unit: participant
Groups:
- Maralixibat (LUM001) 1 mg: Participants received LUM001 tablet orally once daily at a dose of 1 mg during Week 2 of the treatment period.
- Maralixibat (LUM001) 2.5 mg: Participants received LUM001 tablet orally once daily at a dose of 2.5 mg during Week 3 of the treatment period.
- Maralixibat (LUM001) 5 mg: Participants received LUM001 tablet orally once daily at a dose of 5 mg during Week 4 of the treatment period.
- Maralixibat (LUM001) 7.5 mg: Participants received LUM001 tablet orally once daily at a dose of 7.5 mg during Week 5 of the treatment period.
- Maralixibat (LUM001) 10 mg: Participants received LUM001 tablet orally once daily at a dose of 10 mg during Week 6 of the treatment period followed by stable dosing of 10 mg for 8 weeks.
Arm/Group | Maralixibat (LUM001) 1 mg | Maralixibat (LUM001) 2.5 mg | Maralixibat (LUM001) 5 mg | Maralixibat (LUM001) 7.5 mg | Maralixibat (LUM001) 10 mg
Number analyzed (Participants) | 1 | 2 | 2 | 1 | 21
participant | 1 | 2 | 2 | 1 | 19

2. Primary Outcome: Change From Baseline in Fasting Serum Bile Acid Level at Week 14
Description: Serum bile acid levels were evaluated using blood samples collected.
Time Frame: Baseline, Week 14
Population: Modified intent-to-treat (mITT) population included all participants who received at least 1 dose of investigational product and had at least 1 post baseline serum bile acid laboratory assessment.
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | Maralixibat (LUM001)
Number analyzed (Participants) | 27
micromoles per liter
  Baseline | 38.941 (38.6614)
  Change From Baseline | -14.841 (31.3709)
Statistical Analysis 1: Comparison: Maralixibat (LUM001); Analysis was performed to compare baseline and endpoint data; Test type: Superiority or Other; p = 0.0043, Wilcoxon's signed rank test; Mean Difference (Net) = -14.841, 95% CI 2-sided [-27.251 to -2.432], Standard Error of Mean 6.0373

3. Secondary Outcome: Change From Baseline in Liver Enzyme Levels in Serum
Description: Levels of liver enzymes such as Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (ALP) in serum were evaluated.
Time Frame: Baseline, Week 14
Population: mITT population included all participants who received at least 1 dose of investigational product and had at least 1 post baseline serum bile acid laboratory assessment.
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Maralixibat (LUM001)
Number analyzed (Participants) | 27
units per liter (U/L)
  ALT: Baseline | 108.5 (78.95)
  ALT: Change From Baseline | 10.5 (63.07)
  AST: Baseline | 88.3 (43.70)
  AST: Change From Baseline | 11.7 (34.14)
  ALP: Baseline | 471.6 (316.93)
  ALP: Change From Baseline | 36.7 (170.87)

4. Secondary Outcome: Change From Baseline in Bilirubin Levels at Week 14
Description: Total Bilirubin and Direct (Conjugated) Bilirubin levels were evaluated.
Time Frame: Baseline, Week 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Maralixibat (LUM001)
Number analyzed (Participants) | 27
milligram per deciliter (mg/dL)
  Total Bilirubin Level: Baseline | 1.22 (0.775)
  Total Bilirubin Level: Change From Baseline | 0.24 (0.666)
  Conjugated Bilirubin Level: Baseline | 0.60 (0.510)
  Conjugated Bilirubin Level: Change From Baseline | 0.19 (0.450)

5. Secondary Outcome: Change From Baseline in Pruritus as Measured by Adult Itch Reported Outcome (ItchRO) Weekly Sum Score
Description: The Adult ItchRO instrument was completed twice daily using an electronic diary (eDiary). Each morning and evening score had a range from 0-10, with the higher score indicating increasing itch severity. The following was used for assessing the Adult ItchRO daily score: The score which represented the most severe itching for the day (morning or evening) was taken for each day as the daily score (maximum daily score of 10); If only 1 of the 2 scores was available for the day, the score that was available was used as the daily score; If both the morning and the evening scores were missing, the score was considered missing for the day.
Time Frame: Baseline, Week 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Maralixibat (LUM001)
Number analyzed (Participants) | 27
units on scale
  Baseline | 15.00 (18.735)
  Change From Baseline | -7.67 (16.326)

6. Other Pre Specified Outcome: Change From Baseline for Other Biochemical Markers of Cholestasis: Total Cholesterol, Low Density Lipoprotein Cholesterol
Description: Total cholesterol (TC) level and low density lipoprotein cholesterol (LDLC) level were considered as biochemical markers of cholestasis.
Time Frame: Baseline, Week 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Maralixibat (LUM001)
Number analyzed (Participants) | 27
mg/dL
  TC Level: Baseline | 213.0 (50.62)
  TC Level: Change From Baseline | -21.2 (25.46)
  LDLC Level: Baseline | 121.4 (40.52)
  LDLC Level: Change From Baseline | -16.3 (17.64)

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow up (Week 18)
Arm/Group | Maralixibat (LUM001)
Serious Adverse Events (participants affected / at risk) | 4/27
Other Adverse Events (participants affected / at risk) | 25/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maralixibat (LUM001) (N=27)
Melaena (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maralixibat (LUM001) (N=27)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (9)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 3 (4)
Abdominal distension (Gastrointestinal disorders) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 8 (8)
Abdominal pain upper (Gastrointestinal disorders) | 2 (4)
Diarrhoea (Gastrointestinal disorders) | 14 (27)
Frequent bowel movements (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 9 (12)
Asthenia (General disorders) | 2 (2)
Fatigue (General disorders) | 4 (4)
Pyrexia (General disorders) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 2 (2)
Hepatomegaly (Hepatobiliary disorders) | 2 (2)
Headache (Nervous system disorders) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.